CLINICAL TRIAL: NCT05069649
Title: Multicenter, Double-blind, Placebo-controlled, Randomized, Parallel-group Clinical Trial to Evaluate the Efficacy and Safety of Ergoferon as Non-specific COVID-19 Prevention During Vaccination Against SARS-CoV-2
Brief Title: Efficacy and Safety of Ergoferon for COVID-19 Prevention During Vaccination Against SARS-CoV-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MMH-ER-010
Record Dates: First submitted 2021-10-04; First posted 2021-10-06 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2021-11

CONDITIONS: Immunization Against COVID-19
Keywords: Immunization Against COVID-19
MeSH Terms: interventions — ergoferon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ergoferon (Experimental): Tablet for oral use. 1 tablet twice daily. The tablets are taken outside of meals (between meals or 15-30 minutes before meals), keep the tablets in the mouth, without swallowing, until completely dissolved.
  Interventions: Drug: Ergoferon
- Placebo (Placebo Comparator): Tablet for oral use. Placebo using Ergoferon scheme.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ergoferon — Tablet for oral use.
  Arms: Ergoferon
Drug: Placebo — Tablet for oral use.
  Arms: Placebo

SUMMARY:
The multicenter, double-blind, placebo-controlled, parallel-group, randomized clinical trial.

The objective of this study is to evaluate the efficacy and safety of Ergoferon as a non-specific preventive medicine for COVID-19 in individuals vaccinated against a new coronavirus infection (SARS-CoV-2)

DETAILED DESCRIPTION:
Design: the multicenter, double-blind, placebo-controlled, parallel-group, randomized trial.

The study will enroll adult participants of either gender aged ≥18 years who receive a COVID-19 vaccine. The participant signs an information sheet (Informed Consent Form) for participation in the clinical study on the day of administration of component I of the Gam-COVID-Vac (Sputnik-V) vaccine. The physician evaluates if the participant is eligible for the study. A SARS-CoV-2 rapid test (BIOCREDIT COVID-19 Ag) is carried out. If the participant tests positive for SARS-CoV-2, he/she is not enrolled in the study. The investigator's approach should be in compliance with the current version of the guidelines "Prevention, diagnosis, and treatment of a new coronavirus infection (COVID-19)" by the Ministry of Health of the Russian Federation.

If the participant meets all inclusion criteria and does not have any exclusion criteria, then he/she is included in the study, and the physician fills in source medical documentation.

Following enrollment in the study (Day 1, Visit 1), the participant is randomized into one of two groups: participants of the Group 1 receive Ergoferon in the preventive regimen for 3 weeks, and participants of the Group 2 receive Placebo in the same regimen for 3 weeks.

On the day of administration of component II of the Gam-COVID-Vac vaccine (day 22, Visit 2 + 3 days) the express test for SARS-CoV-2 (BIOCREDIT COVID-19 Ag) is performed.

After the component II of the vaccine has been administered, the participant is followed up for 2 weeks. After 2 weeks, Visit 3 ("phone visit") is carried out in order to interview the participant about the health status (absence/presence of any ARVI symptoms).

All participants are provided with classic thermometers for measuring axillary temperature. Electronic diaries are used in the trial to record any potential deterioration in the participant's condition (if applicable) for the assessment of efficacy, safety, and registration of adverse events. The investigator trains the participant how to fill in the diary. Once a week, the participant receives an SMS reminder: "If you have symptoms of the disease, note them in your diary. The investigator will contact you".

If the participant develops symptoms of an acute respiratory viral infection (ARVI)? including an increase in body temperature to febrile/subfebrile values, weakness, headache, chills, cough, sore throat, other symptoms, etc. within five weeks of the observation, the investigator will perform an unscheduled visit to collect nasopharynx and oropharynx swabs for the RT-PCR test (performing in the central laboratory).

If the participant without ARVI symptoms will have a positive test for SARS-CoV-2 (rapid test) at Visit 1 or 2, his/her nasal and oropharyngeal swabs will also be collected for RT-PCR testing in the central laboratory.

If a laboratory-confirmed SARS-CoV-2 infection (with or without symptoms) is detected, the participant will complete the participation in the trial as meeting the primary endpoint.

In case of a positive PCR for SARS-CoV-2, in accordance with the requirements of Rospotrebnadzor Agency, the information about it should be transferred to the medical facility where the participant is registered and where appropriate medical care will be provided for the participant in accordance with the current standards. The employees of the medical facility will report COVID-19 data in compliance with the requirements of the Ministry of Health of the Russian Federation and the rules of the medical facility.

Possible post-vaccination symptoms;

* general (a flu-like syndrome characterized by chills, fever, arthralgia, myalgia, asthenia, general malaise, headache) and local (pain at the injection site, hyperemia, swelling) reactions that develop on the first-second day and resolve within three subsequent days;
* nausea, dyspepsia, loss of appetite;
* enlarged regional lymph nodes;
* allergic reactions;
* short-term increase in serum levels of liver transaminases, creatinine, and creatine phosphokinase.

These post-vaccination symptoms are not recorded as adverse events (either associated with the investigational product administration or developing after discontinuation); they are registered by the participant in the diary and assessed by the physician as post-vaccination complications.

The short-term flu-like syndrome should not be diagnosed as ARVI, in this case, the RT-PCR test for SARS-CoV-2 is not performed.

If the participant is ill with COVID-19 or has been hospitalized for COVID-19, a delayed "phone" visit is performed. The visit is scheduled by the investigator depending on each case.

During the study participants are allowed to take medications for their chronic conditions, except for medicines listed as "Prohibited concomitant treatment".

ELIGIBILITY:
Inclusion Criteria:

1. Adults of either gender aged ≥18 years.
2. Participant has not had COVID-19 in the previous 6 months.
3. The participant has not been vaccinated against COVID-19 or other viral infections in the previous 6 months.
4. Negative rapid test result for SARS-CoV-2 (COVID-19 Ag).
5. Absence of clinical manifestations of any infectious disease, but not earlier than 14 days from its onset.
6. Consent to use reliable contraceptive methods during the study (for men and women with reproductive potential).
7. Presence of a signed information sheet and informed consent form for participation in a clinical trial.

Exclusion Criteria:

1. The presence of contraindications to vaccination:

   * hypersensitivity to any component of the vaccine or a vaccine containing similar components;
   * prior history of severe allergic reactions;
   * acute infectious and non-infectious diseases, exacerbation of chronic diseases.
2. Severe chronic hepatic and renal disorders, severe thyroid dysfunction, decompensated diabetes mellitus, severe disorders of the hematopoietic system, epilepsy and other CNS diseases, acute coronary syndrome, acute cerebrovascular accident, myocarditis, endocarditis, pericarditis, autoimmune diseases, or immunodeficiency.
3. Malabsorption syndrome, including congenital or acquired lactase deficiency or any other disaccharidase deficiency, galactosemia.
4. Hypersensitivity to any of the components of study drug used in the treatment.
5. Pregnancy, breast-feeding, childbirth less than 3 months before study enrollment.
6. Participants who, from the investigator's point of view, will not comply with study observation requirements or study drug administration procedures.
7. Inability to observe the participant during the study period.
8. Prior history of mental illness, alcoholism or drug abuse, that the investigator's opinion, will interfere with successful study procedures.
9. Participation in other clinical studies within 3 months prior to enrollment in the study.
10. Use of any medications listed in "Prohibited concomitant treatment" within 4 weeks before enrollment.
11. Participants who are related to any of the on-site research personnel directly involved in the conduct of the trial or are an immediate relative of the study investigator. "Immediate relative" means husband, wife, parent, son, daughter, brother, or sister (regardless of whether they are natural or adopted).
12. Participants who work for OOO "NPF "MATERIA MEDICA HOLDING" (i.e. the company's employees, temporary contract workers, designated officials responsible for carrying out the research or any immediate relatives of the aforementioned).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1057 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- Russia (32):
  - Belgorod State National Research University, Department of Hospital Therapy, Belgorod
  - City Clinical Hospital # 9 of the Ministry of Health of the Udmurt Republic, Izhevsk
  - Baltic Federal University named after Immanuel Kant, Kaliningrad
  - Kazan State Medical University/Department of Internal Diseases, Kazan'
  - Republican Clinical Infectious Diseases Hospital named after Prof. A.F. Agafonov, Kazan'
  - Kirov State Medical University, Hospital Therapy Department, Kirov
  - Specialized Clinical Infectious Diseases Hospital/Vaccination room, Krasnodar
  - Kuban State Medical University, Infectious Diseases and Phthisiopulmonology, Krasnodar
  - Central Clinical Hospital of the Russian Academy of Sciences, Moscow
  - Llc "Verum Medical", Moscow
  - Road Clinical Hospital at the station Nizhny Novgorod of JSC Russian Railways, Nizhny Novgorod
  - Clinical Hospital # 4, Penza
  - City Emergency Hospital of Rostov-on-Don, Rostov-on-Don
  - LLC "BioTechService", Saint Petersburg
  - LLC "Research Center Eco-safety", Saint Petersburg
  - City Polyclinic # 25 of the Nevsky District, Saint Petersburg
  - LLC "Energy of Health", Saint Petersburg
  - LLC "Clinic Zvezdnaya", Saint Petersburg
  - City Polyclinic # 51, Saint Petersburg
  - City Polyclinic # 34, Saint Petersburg
  - City polyclinic #106, Saint Petersburg
  - LLC "Meili", Saint Petersburg
  - City polyclinic # 74, Saint Petersburg
  - Samara City Hospital # 4, Samara
  - LLC "DNA Research Center", Saratov
  - Saratov State Medical University named after V. I. Razumovsky, Saratov
  - LLC "Scientific Medical Center for General Therapy and Pharmacology", Stavropol
  - Bashkir State Medical University, Internal Medicine Department, Ufa
  - Clinical Hospital # 2/Therapeutic department, Yaroslavl
  - Central City Hospital, Yaroslavl
  - Clinical Hospital # 9/Polyclinic #1, Yaroslavl
  - Central City Hospital # 7, Yekaterinburg

REFERENCES:
- [Derived] Avdeeva MG, Belousova ON, Orlova EA, Khamitov RF, Shvarts YG, Kravchenko IE. [Non-specific prevention of COVID-19 during vaccination against a new coronavirus infection: results of a multicenter, double-blind, placebo-controlled, randomized clinical trial]. Ter Arkh. 2022 Dec 26;94(11):1268-1277. doi: 10.26442/00403660.2022.11.201980. Russian. PMID 37167165

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 participants were not screened because they did not meet the inclusion / non-inclusion criteria.
Period: Overall Study
Arm/Group | Ergoferon | Placebo
Started | 526 | 524
Completed | 526 | 524
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ergoferon | Placebo | Total
Number analyzed (Participants) | 526 | 524 | 1050
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 439 | 439 | 878
  >=65 years | 87 | 85 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (17.2) | 45.0 (17.0) | 45.2 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 291 | 278 | 569
  Male | 235 | 246 | 481
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 526 | 524 | 1050

OUTCOME MEASURES:

1. Primary Outcome: The Number of Laboratory-confirmed SARS-CoV-2 Infections.
Description: Based on medical records. The number of laboratory-confirmed SARS-CoV-2 infections (with or without symptoms) in vaccinated individuals throughout the trial. A laboratory-confirmed case will be defined as a case where the novel SARS-CoV-2 coronavirus is detected by RT-PCR in a symptomatic or asymptomatic participant with COVID-19.
Time Frame: 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 526 | 524
Participants | 7 | 22
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; Test type: Superiority; p = 0.0046, Chi-squared

2. Secondary Outcome: The Percentage of Hospitalized Participants With COVID-19.
Description: Based on medical records.
Time Frame: 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 526 | 524
Participants | 0 | 2
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; Test type: Superiority; p = 0.2488, Fisher Exact

3. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: The presence and nature of AEs. Based on medical records.
Time Frame: 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 526 | 524
Participants | 15 | 15
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; Test type: Superiority; p = 1.0, Fisher Exact

4. Secondary Outcome: Severity of AEs
Description: The intensity (severity) and outcomes of adverse events. Mild - AE allows you to perform everyday activities and does not require treatment; Moderate - AE interferes with daily activities and/or requires treatment; Severe - AE makes it impossible to perform daily activities and/or requires the appointment of therapy.
  Based on medical records.
Time Frame: 3 weeks
Measure: Number; unit: number of AE
Units Other Than Participants: Adverse Events (AEs)
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 526 | 524
Number analyzed (Adverse Events (AEs)) | 19 | 20
number of AE
  Mild | 13 | 11
  Moderate | 5 | 9
  Severe | 1 | 0
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; Test type: Superiority; p = 0.32, Fisher Exact

5. Secondary Outcome: Causal Relationship of AEs to the Sudy Drug
Description: The causal relationship to the study drug of adverse events. Based on medical records.
Time Frame: 3 weeks
Measure: Number; unit: number of AE
Units Other Than Participants: Adverse Events (AEs)
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 526 | 524
Number analyzed (Adverse Events (AEs)) | 19 | 20
number of AE
  No relation | 14 | 20
  Possible | 1 | 0
  Doubtful | 3 | 0
  Сonventional | 1 | 0
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; Test type: Superiority; p = 0.02, Fisher Exact

6. Secondary Outcome: Outcome of AEs
Description: The outcome of adverse events. Based on medical records.
Time Frame: 3 weeks
Measure: Number; unit: number of AE
Units Other Than Participants: Adverse Events (AEs)
Arm/Group | Ergoferon | Placebo
Number analyzed (Participants) | 526 | 524
Number analyzed (Adverse Events (AEs)) | 19 | 20
number of AE
  Recovery/resolution | 18 | 20
  Incomplete recovery/ resolution | 1 | 0
Statistical Analysis 1: Comparison: Ergoferon vs Placebo; Test type: Superiority; p = 0.49, Fisher Exact

ADVERSE EVENTS:
Time Frame: Registration of AEs begins after taking the first dose of study drug and continues throughout the entire period of patient's participation in the study - 3 weeks.
Arm/Group | Ergoferon | Placebo
All-Cause Mortality (participants affected / at risk) | 0/526 | 0/524
Serious Adverse Events (participants affected / at risk) | 1/526 | 0/524
Other Adverse Events (participants affected / at risk) | 15/526 | 15/524
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ergoferon (N=526) | Placebo (N=524)
Bradycardia-tachycardia syndrome (Cardiac disorders) | 1 (1) | 0 (0) — Sick sinus syndrome. Tachy-Brady syndrome. Sinus bradycardia. Hospitalization. Emergency pacemaker implanted. Incomplete recovery.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ergoferon (N=526) | Placebo (N=524)
Acute gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Digestive disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Viral respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia of the right middle lobe (Infections and infestations) | 1 (1) | 0 (0)
Rhinosinusitis (Infections and infestations) | 0 (0) | 1 (1)
Increased blood pressure (Investigations) | 2 (2) | 4 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Non-infectious rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Exertional dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Post-vaccination reaction (Immune system disorders) | 0 (0) | 1 (1)
Brachialgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 5 (5)
Migraine (Nervous system disorders) | 2 (2) | 0 (0)
Injection site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
General weakness (General disorders) | 1 (1) | 0 (0)
Precardial pain (General disorders) | 0 (0) | 1 (1)
Weakness (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT05069649/Prot_SAP_000.pdf